CLINICAL TRIAL: NCT05973747
Title: Pharmacokinetic Equivalence of Calcium Gluconate and Calcium Chloride in Parturients
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Jessica Ansari, MD, Clinical Assistant Professor of Anesthesiology, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 70603
Record Dates: First submitted 2023-07-13; First posted 2023-08-03 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Postpartum Hemorrhage; Pregnancy Related; Hypocalcemia; Parturition Complication
MeSH Terms: conditions — Postpartum Hemorrhage; Hypocalcemia | interventions — Calcium Gluconate; Calcium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Calcium Gluconate (Experimental): Infused intravenously over 10 minutes upon umbilical cord clamping. First 10 assigned patients received 2 grams per protocol. Subsequent 13 patients received 1.5 grams, dose recalibrated per protocol.
  Interventions: Drug: Calcium Gluconate
- Calcium Chloride (Active Comparator): 0.5mg calcium chloride, infused intravenously over 10 minute infusion beginning upon umbilical cord clamping
  Interventions: Drug: Calcium chloride

INTERVENTIONS:
Drug: Calcium Gluconate — Infused intravenously over 10 minutes upon umbilical cord clamping. First 10 assigned patients received 2 grams per protocol. Subsequent 13 patients received 1.5 grams, dose recalibrated per protocol.
  Arms: Calcium Gluconate
Drug: Calcium chloride — 0.5 grams of calcium chloride, infused intravenously over 10 minutes upon umbilical cord clamping
  Arms: Calcium Chloride

SUMMARY:
Calcium is a life saving medicine in the care of parturients. It has many important uses including treatment of hypocalcemia, treatment of magnesium toxicity, prevention of hypocalcemia during blood transfusion (of citrate containing blood products), treatment of hyperkalemia, and others. Recent clinical trials also suggest that calcium given after cord clamping may decrease blood loss in patients undergoing cesarean delivery. 2 FDA approved forms of calcium can be given intravenously: calcium chloride and calcium gluconate. Over the last decade there have been times with drug shortages of either calcium chloride or calcium gluconate. So there have been and likely will continue to be times when one formulation or the other may not be adequately available. Despite the importance of calcium and the frequency in which it is used in parturients, there are no published studies in parturients to determine dose equivalence between calcium gluconate and calcium chloride. In this study the investigators will determine the population pharmacokinetics of calcium gluconate and calcium chloride in parturients and calculate the dose equivalent ratio the two drugs. This will help clinicians select appropriate doses of calcium and provide resilience to the drug supply chain in our era of frequent drug shortages.

ELIGIBILITY:
Inclusion Criteria:

Pregnant female subjects delivering at the study institution via scheduled cesarean delivery at term (>=37 weeks gestation)

Exclusion Criteria:

1. severe range blood pressure (BP >160/>110) within the 48 hours prior to delivery
2. patient age <18 years or >45 years
3. renal dysfunction with serum Cr > 1.0 mg/dL
4. known history of congenital or acquired cardiac disease or history of arrhythmia
5. patient taking digoxin
6. patient currently taking a calcium channel blocker
7. Weight <55kg or >100kg, or
8. receiving magnesium infusion within 24 hours prior to or during cesarean delivery
9. administration of intraoperative doses of calcium by the anesthesiology team for clinical indications

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Parturients all biologically female at birth by necessity
Enrollment: 34 (Actual)
Dates: Start 2023-08-19 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Bioequivalent ratio of calcium gluconate (g) to calcium chloride (g) | Using data gathered from serial lab draws at 5 minutes, 10 minutes, 15 minutes, 30 minutes, 60 minutes after initiation of infusion
  Calculated via NONMEM
Clearance from first to second compartment (L/min) | Using data gathered from serial lab draws at 5 minutes, 10 minutes, 15 minutes, 30 minutes, 60 minutes after initiation of infusion
  Determined using population pharmacokinetic analysis in NONMEM
Volume of distribution of first compartment of pharmacokinetic model (L) | Using data gathered from serial lab draws at 5 minutes, 10 minutes, 15 minutes, 30 minutes, 60 minutes after initiation of infusion
  Determined using population pharmacokinetic analysis in NONMEM
Clearance from second compartment (L/min) | Using data gathered from serial lab draws at 5 minutes, 10 minutes, 15 minutes, 30 minutes, 60 minutes after initiation of infusion
  Determined using population pharmacokinetic analysis in NONMEM
Volume of distribution of second compartment of pharmacokinetic model (L) | Using data gathered from serial lab draws at 5 minutes, 10 minutes, 15 minutes, 30 minutes, 60 minutes after initiation of infusion
  Determined using population pharmacokinetic analysis in NONMEM

SECONDARY OUTCOMES:
Serum pH | Baseline prior to calcium infusion, 6 minutes, 10 minutes, 15 minutes, 30 minutes, 60 minutes after initiation of infusion
  Serum pH will be measured in each participant from a maximum of 6 venous blood draws of 0.5mL (1/10th of a teaspoon). These blood draws will be the same blood draws used to measure serum ionized calcium concentration, no additional blood draws will be necessary. These draws will occur at the following target times: prior to calcium administration, at 6 minutes, 10 minutes, 15 minutes, minutes, minutes after beginning calcium administration. The serum pH levels will be immediately analyzed using an Abbott iStat machine.
Baseline serum ionized calcium concentration | Baseline prior to calcium infusion
  Ionized calcium will be measured in each participant prior to administration of the 10-minute calcium infusion. The ionized blood calcium levels will be immediately analyzed using an Abbott iStat machine.
Peak change in serum ionized calcium concentration (mmol/L) | Measured immediately at completion of the 10-minute calcium infusion.
  Measured via venous blood draw and an Abbott iStat CG8+ cartridge
Time to half of peak change in ionized calcium (minutes) | 10-60 minutes after infusion initiation
  A two-compartment model does not lend itself to a meaningful half-life approximation. However, the time to serum values measuring 1/2 of the peak change in ionized calcium can be calculated from the pharmacokinetic model

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Ansari, MD, MS, Principal Investigator — Stanford University
Locations (1):
- Lucile Packard Children's Hospital, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No